CLINICAL TRIAL: NCT04112316
Title: Developing Oral LT3 Therapy For Heart Failure With Reduced Ejection Fraction
Brief Title: Developing Oral LT3 Therapy for Heart Failure - HFrEF
Acronym: DOT3HF-HFrEF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Anne Cappola, MD, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 833681r; 1R61HL146390-01 (NIH)
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF); Low T3 Syndrome
Keywords: Heart Failure; HFrEF; Low T3 Syndrome
MeSH Terms: conditions — Euthyroid Sick Syndromes; Heart Failure | interventions — Triiodothyronine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant, Investigators and Care Providers are blinded to LT3 vs. Placebo and T3 results. There will be 1 unblinded physician in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liothyronine (LT3), then placebo (Active Comparator): Participants received liothyronine first, with weekly titration of study drug for four weeks, followed by a maintenance dose for 4 weeks, then 2-week washout before crossing over to receive placebo for 8 weeks.
  Interventions: Drug: Liothyronine; Other: Placebo
- Placebo, then liothyronine (Placebo Comparator): Participants received placebo first, with weekly sham titration for four weeks, followed by a maintenance dose for 4 weeks, then 2-week washout before crossing over to receive LT3 for 8 weeks.
  Interventions: Drug: Liothyronine; Other: Placebo

INTERVENTIONS:
Drug: Liothyronine — Liothyronine (L-triiodothyronine or LT3) in the 5 mcg tablet dose formulation. Minimum LT3 dose was 2.5 mcg three times daily and the maximum LT3 dose was 12.5 mcg three times daily.
  Other Names: LT3
Other: Placebo — A placebo tablet matching in appearance to LT3 tablets. Minimum placebo tablet dose was 1/2 tablet three times daily and the maximum placebo dose was 2 1/2 tablets three times daily.

SUMMARY:
Investigation of the safety, feasibility, and preliminary efficacy of thyroid hormone therapy with Liothyronine (LT3) in individuals with heart failure with reduced ejection fraction (HFrEF) and low triiodothyronine (T3) syndrome by conducting a randomized, double-blind, placebo-controlled cross-over study with a two-week washout period between treatments.

DETAILED DESCRIPTION:
The overall goal is to determine the safety, feasibility, and preliminary efficacy of administering oral LT3 therapy in the study population of participants with Heart Failure with reduced ejection fraction (HFrEF). The study will consist of two treatment periods - each treatment period will be approximately 8 weeks in duration, with weekly titration of study drug for 4 weeks, followed by a maintenance dose for 4 weeks, then 2-week washout before crossing over to the other arm (placebo or drug). LT3 will be titrated to T3 levels.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥18 years
2. NYHA Class I, II or III heart failure
3. EF≤40 percent within the past year
4. An implantable cardioverter-defibrillator (ICD)
5. Stable doses of neurohormonal blockade for 30 days
6. TSH and free T4 level within the laboratory reference range and total T3 level <94 ng/dL

Exclusion Criteria:

1. Hypertrophic or restrictive cardiomyopathy
2. Uncorrected severe primary valvular disease
3. Arrhythmia that results in irregular heart rate
4. Inability to perform VO2max exercise testing
5. Severe lung disease, including treatment with oral steroids within past 6 months for exacerbation of obstructive lung disease or use of daytime supplemental oxygen
6. Serum creatinine > 3.0 mg/dL
7. History of cirrhosis
8. LVAD use
9. Heart failure hospitalization within past month
10. Acute coronary syndrome, coronary intervention or ablation therapy within past 2 months or cardiac surgery, percutaneous repair of a valve or septal defect repair within the past 6 months
11. Taking thyroid extract, LT4, LT3, amiodarone, or medication that affects the absorption or metabolism of thyroid hormone; gastrointestinal conditions that affect the absorption of thyroid hormone
12. If female, current or planned pregnancy within the timeframe of study participation
13. Any medical condition that in the opinion of the investigator, will interfere with the safe completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne R Cappola, MD,ScM, Principal Investigator — University of Pennsylvania
Locations (1):
- PennMedicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Period (8 Weeks)
Arm/Group | Liothyronine (LT3), Then Placebo | Placebo, Then Liothyronine
Started | 14 | 14
Completed | 12 | 14
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Washout (2 Weeks)
Arm/Group | Liothyronine (LT3), Then Placebo | Placebo, Then Liothyronine
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0
Period: Second Intervention (8 Weeks)
Arm/Group | Liothyronine (LT3), Then Placebo | Placebo, Then Liothyronine
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liothyronine (LT3), Then Placebo | Placebo, Then Liothyronine | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 8 | 13
  >=65 years | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (11.0) | 59.0 (12.3) | 61.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 12 | 14 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Rhythm Monitoring by 14 Day Patch Rhythm Assessment
Description: Number of participants with atrial fibrillation or ventricular tachycardia >= 4 beats
Time Frame: continuous during intervention (14 days)
Measure: Number; unit: Number of participants with events
Groups:
- Liothyronine (LT3): Participants who received liothyronine for the first 8 weeks or the last 8 weeks of the study.
- Placebo: Participants who received placebo for the first 8 weeks or the last 8 weeks of the study.
Arm/Group | Liothyronine (LT3) | Placebo
Number analyzed (Participants) | 28 | 26
Number of participants with events | 11 | 19

2. Primary Outcome: T3 Level
Description: Number of participants with T3 levels above upper limit of reference range
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Liothyronine (LT3) | Placebo
Number analyzed (Participants) | 26 | 26
Participants | 4 | 0

3. Secondary Outcome: Change in Peak Maximal Rate of Oxygen Consumption During Exercise (VO2 Max)
Description: Change in peak rate of oxygen consumption during exercise between baseline and 8 weeks
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Liothyronine (LT3) | Placebo
Number analyzed (Participants) | 23 | 23
ml/kg/min | 11.18 (4.24) | 10.78 (4.31)

4. Secondary Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Quality of Life
Description: Change in KCCQ from baseline to 8 weeks, 0-100 scale, higher is better
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liothyronine (LT3) | Placebo
Number analyzed (Participants) | 27 | 26
units on a scale | 0.6 (6.8) | -0.6 (10.3)

5. Secondary Outcome: Activity Measured Via Actigraphy
Description: Remotely sensed minutes/day of cumulative light, moderate, or vigorous activity in minutes/day after 8 weeks of LT3 or placebo
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Liothyronine (LT3) | Placebo
Number analyzed (Participants) | 23 | 23
minutes/day | 241 (83) | 265 (82)

6. Secondary Outcome: Change in NT-proBNP Levels
Description: Change in B-type natriuretic peptide levels, Pg/mL, from baseline to 8 weeks
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Liothyronine (LT3) | Placebo
Number analyzed (Participants) | 26 | 26
pg/mL | 66.1 (248.3) | 98.7 (450.9)

ADVERSE EVENTS:
Time Frame: 17 weeks
Arm/Group | Liothyronine (LT3) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 15/28 | 9/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liothyronine (LT3) (N=28) | Placebo (N=28)
Total (Investigations) | 15 (25) | 9 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT04112316/Prot_SAP_000.pdf